CLINICAL TRIAL: NCT05100966
Title: Getting Fit for Hip and Knee Replacement: The FitJoints Multisite Randomized Controlled Trial of a Multi-modal Intervention in Frail Patients With Osteoarthritis
Brief Title: FitJoints: Getting Fit for Hip and Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); St. Joseph's Health Care London (Other); London Health Sciences Centre (Other); Alberta Health services (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Professor, Department of Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3732
Record Dates: First submitted 2021-09-27; First posted 2021-10-29 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: Frail elderly; Arthroplasty; Pre-rehabilitation
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants in the control arm will receive usual care which involves patient education that all participants who are scheduled for hip/knee replacement receive at the arthroplasty centre. This may include recommendations to attend fitness classes or discuss nutrition tips and smoking cessation initiatives with their family doctor or other healthcare provider before surgery.
- FitJoints Multi-modal Intervention (Active Comparator)
  Interventions: Other: FitJoints Multi-modal Intervention

INTERVENTIONS:
Other: FitJoints Multi-modal Intervention — Exercise: The study physiotherapist will prescribe an exercise program tailored to the participant's individual ability and preference with functional movements to mimic activities of daily living.
  Nutritional consultation and protein supplement: The site research assistant will coach participants to improve their nutrition, determine their daily protein target, and provide educational tools on how to achieve their target. Protein supplements will be provided to participants.
  Vitamin D: Participants will be provided with vitamin D3 (1000 IU) tablets to reduce the risk of falls and to preserve muscle strength and functional ability. They will be instructed to take one tablet daily for the duration of the intervention period.
  Medication optimization: The study pharmacist will conduct a medication review and provide, if required, recommendations for medication optimization.
  Arms: FitJoints Multi-modal Intervention

SUMMARY:
Total hip or knee replacement is an important and cost-effective surgical intervention to relieve pain and improve independence and function in patients with osteoarthritis. The number of people waiting for elective surgeries has spiked in the COVID-19 pandemic. Prior to COVID-19, up to 40% of patients receiving joint replacement were frail and this number is rapidly increasing with longer wait-times and deconditioning associated with COVID-19 physical distancing. There is an urgent need to be responsive to the evolving challenges of healthcare. The proposed study is the first multi-site randomized controlled trial (RCT) to examine whether a multimodal frailty reduction intervention before surgery will improve postsurgical outcomes for this population. The COVID-19 adapted hybrid model includes a multimodal frailty intervention that may be implemented either in person or virtually and is aligned with international consensus guidelines on frailty reduction.

To utilize the FitJoints multimodal frailty intervention to build resilience of patients undergoing joint replacement surgery to improve post-operative outcomes. The investigators hypothesize the FitJoints multimodal frailty intervention, with exercise, nutrition and medication optimization, will reduce frailty and pain while improving function and quality of life.

Building upon the success of the FitJoints feasibility study (n=69) in Hamilton, Ontario, in the proposed multi-site RCT (n=192), older adults (≥60 years) undergoing hip or knee joint replacement surgery who are frail will be randomized to either the 3 to 6-months of multimodal intervention or usual care until the date of their surgery at multiple sites (Hamilton Health Sciences & St Joseph's Healthcare Hamilton, ON; London Health Science Centre, London, ON; Foothills Hospital, Calgary, AB),The FitJoints evidence-based, multimodal intervention includes a hybrid model that can be implemented either in person or virtually:

1. Physiotherapist supported multi-component exercise program
2. Nutrition and protein optimization including dietary counseling
3. Medication review with prescribing recommendations

ELIGIBILITY:
Inclusion Criteria:

* Pre-frail (score of 1 or 2) or frail (score of 3-5)
* ≥ 60 years old
* Receiving elective unilateral total hip or knee replacement
* Waiting time for surgery is estimated to be between 4 to 15 months

Exclusion Criteria:

* Renal disorder
* A neuromuscular disorder
* Active cancer
* Inflammatory arthritis
* Unable to speak or understand English and has no caregiver for translation
* Participating in another trial that involves protein supplementation
* Participating in an exercise program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Between-group Difference in Physical Performance | 3-months post-operative
  Assessed by the Short Physical Performance Battery (SPPB), which consists of the following sub-components:
  * 4-meter walk test (walking speed): measured in seconds, scored 0 to 4
  * Chair rise: the ability to rise from a chair without arms: measured in seconds, scored 0 to 4
  * Standing balance test: measured in seconds, scored 0 to 4
  Sub-component scores will be aggregated to produce an overall SPPB score, with higher scores indicating lower level of frailty [range 0-12].

SECONDARY OUTCOMES:
Between-group Difference in Frailty | 3-months post-operative
  Assessed by the Fit-Frailty Index. Higher scores indicate greater degree of frailty [range 0-1].
Between-group Difference in Knee Function/Pain | 3-months post-operative
  Patient-reported knee function/pain, assessed by the Oxford Knee Score. Higher scores indicate better knee functionality [range 0-48].
Between-group Difference in Hip Function/Pain | 3-months post-operative
  Patient-reported hip function/pain, assessed by the Oxford Hip Score. Higher scores indicate better hip functionality [range 0-48].
Between-Group Difference in Instrumental Activities of Daily Living | 3-months post-operative
  Ability to carry out instrumental activities of daily living as operationalized by the Older American Resources & Services (OARS) questionnaire. Higher scores indicate greater ability to perform instrumental activities of daily living [range 0-14].
Between-group Difference in Physical Activities of Daily Living | 3-months post-operative
  Ability to carry out physical activities of daily living as operationalized by the Older American Resources & Services (OARS) questionnaire. Higher scores indicate greater ability to perform physical activities of daily living [range 0-14].
Between-group difference in Sarcopenia | 3-months post-operative
  Assessed by the SARC-F - Self-reported strength, assistance with walking, rising from a chair, climbing stairs and falls. Higher scores indicate greater level of sarcopenia, with scores equal to or greater than 4 predictive of sarcopenia and poorer outcomes [range 0-10].
Between-group Difference in Nutrition | 3-months post-operative
  Assessed by the Mini Nutritional Assessment (MNA). Higher scores indicate better nutritional status (<17 malnourished, 17-23.5 at risk of malnutrition, 24-30 normal nutritional status) [range 0-30].
Between-group Difference in Cognition | 3-months post-operative
  Ottawa-3DY-cognitive assessment - recall of day of week, date, year, spell WORLD backwards. Score of 4 indicates normal mental status, <4 indicates impaired mental status [range 0-4].
Between-group Difference in Health-Related Quality of Life | 3-months post-operative
  Quality of life questionnaire (EQ-5D-5L) which consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Between-group Difference in Number of Hospitalizations | 3-months post-operative
  Number of hospitalizations will be recorded. Higher numbers of hospitalizations indicates higher healthcare utilization.
Between-group Difference in Number of Emergency Department Visits | 3-months post-operative
  Number of emergency department visits will be recorded. Higher number of emergency department visits indicates higher healthcare utilization.
Between-group Difference in Number of Visits to Physicians/Healthcare Professionals | 3-months post-operative
  Number of visits to physicians and other healthcare professionals will be recorded. Higher number of visits indicates higher healthcare utilization.
Between-group Difference in Number of Post-operative Complications | 3-months post-operative
  Any post-op complications (e.g. number of infections, peri-prosthetic fractures, bleeding) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Foothill Medical Centre - Alberta Health Services, Calgary, Alberta
  - Juravinski Hospital - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - University Hospital - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No